CLINICAL TRIAL: NCT00753402
Title: The Effects of Epinephrine in Endotoxemia in Normal Volunteers
Acronym: Epi
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 0220003283
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Immune System
MeSH Terms: interventions — Endotoxins; Lipopolysaccharides; Sodium Chloride; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): IV Endotoxin plus saline vehicle (placebo)
  Interventions: Biological: Endotoxin, Lipopolysaccharide, LPS
- B (Active Comparator): IV Endotoxin plus IV epinephrine
  Interventions: Biological: Endotoxin, Lipopolysaccharide, LPS; Biological: Endotoxin, Epinephrine

INTERVENTIONS:
Biological: Endotoxin, Lipopolysaccharide, LPS — Clinical Center Reference Endotoxin, lot 2, sterile saline, 2 ng/kg, bolus IV administration (~5 minutes)
  Other Names: Sodium Chloride Solution
Biological: Endotoxin, Epinephrine — Clinical Center Reference Endotoxin, lot 2, sterile saline, 2 ng/kg, bolus IV administration (~5 minutes/Epinephrine 30mcg/kg/min
  Other Names: Adrenaline Chloride
  Arms: B

SUMMARY:
Epinephrine (adrenaline) is a substance produced by the body (in the adrenal gland) in response to stress such as infection or injury. Endotoxin is a man- made substance, which causes the body to "mimic" sickness (fever, chills, and achiness) for a few hours. This study is designed to give epinephrine before and/or after endotoxin to determine if this medication can prevent or relieve any of the symptoms caused by endotoxin.

DETAILED DESCRIPTION:
The body's immune response to injury otr infection is very complex. immune cell activity, the release of specific mediators (such as proteins), genetics (Deoxyribonucleic acid or DNA) and/or the body's "instructions" for making proteins (Ribonucleic Acid or RNA) may effect the body's clinical response to a stress such as an infection.Epinephrine (adrenaline) is a substance produced by the body (in the adrenal gland)in response to stress such as infection or injury. Endotoxin is a man- made substance, which causes the body to "mimic" sickness (fever, chills, and achiness) for a few hours. This study is designed to give epinephrine before and/or after endotoxin to determine if this medication can prevent or relieve any of the symptoms caused by endotoxin.In addition, this study may determine whether any of the above(proteins,DNA,RNA,etc.) correlate with or affect the body's response to epinephrine and/or endotoxin. This will enable the investigator to better understand whether treatment with this substance can alter the body's immune response.

ELIGIBILITY:
Inclusion Criteria:

* General good health as demonstrated by medical history, physical& laboratory tests
* Age between 18 and 40 years
* Written informed consent prior to the performance of any study related procedures

Exclusion Criteria:

* History of cancer, rheumatoid arthritis, or immunological, renal, hepatic, endocrine, neurologic, heart disease or hypertension
* Any medication taken in past 48 hrs (except birth control)
* Recent history of alcohol or drug abuse
* Unable to provide written informed consent
* Exposure to any experimental agent or procedure within 30 days of study
* Pregnant or breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Physiological, Hematological, Immunological Responses | 0.5-24 hrs post Endotoxin administration

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan Corbett, MD, Principal Investigator — Rutgers-RWJMS
Locations (1):
- Rutgers-RWJMS, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Matot I, Paskaleva R, Eid L, Cohen K, Khalaileh A, Elazary R, Keidar A. Effect of the volume of fluids administered on intraoperative oliguria in laparoscopic bariatric surgery: a randomized controlled trial. Arch Surg. 2012 Mar;147(3):228-34. doi: 10.1001/archsurg.2011.308. Epub 2011 Nov 21. PMID 22106246
- [Derived] Jan BU, Coyle SM, Oikawa LO, Lu SE, Calvano SE, Lehrer PM, Lowry SF. Influence of acute epinephrine infusion on endotoxin-induced parameters of heart rate variability: a randomized controlled trial. Ann Surg. 2009 May;249(5):750-6. doi: 10.1097/SLA.0b013e3181a40193. PMID 19387330